CLINICAL TRIAL: NCT01868113
Title: Acute Respiratory Infections and Asthma in U-5 Children: Improved Treatment to Reduce Morbidity and Mortality in Uganda, A Randomized Controlled Trial
Brief Title: Inhaled Corticosteroids in U-5 Children With Acute Respiratory Infection in Uganda: A Randomised Trial
Acronym: ICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HS1259
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-04

CONDITIONS: Bacterial Pneumonia; Viral Pneumonia; Acute Asthma
Keywords: Children U-5; ALRI; Inhaled Corticosteroids
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumonia, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled fluticasone propionate (Active Comparator): Inhaled corticosteroid
  Interventions: Drug: Inhaled corticosteroid
- Inhaler propellant (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Inhaled corticosteroid — Inhaled fluticasone 500mcg 12 hourly up to discharge or a maximum of 5 days
  Other Names: Inhaled fluticasone propionate
  Arms: Inhaled fluticasone propionate
Other: Placebo — Placebo to be administered 12hourly
  Other Names: Inhaler propellant
  Arms: Inhaler propellant

SUMMARY:
The purpose of this study is to find out whether adjunct treatment with inhaled corticosteroids lead to faster improvement and reduce mortality of children under 5 years of age admitted to hospital with ALRI.

DETAILED DESCRIPTION:
Pneumonia is one of the common causes of serious illness in children under 5 years of age. It is one of the common causes of admission to hospital and the commonest cause of death in Ugandan children under 5 years of age. The signs of pneumonia also occur in children with asthma making it difficult to differentiate the two. Other researchers have found that one of two children under five years of age with pneumonia have asthma. Wheeze which is regarded as a sign of asthma is heard in only one of three children with asthma, implying that many children with asthma especially in the first few years of life are less likely to be diagnosed. They are also less likely to receive inhaled steroids, the recommended treatment for asthma. Failure to administer asthma medicines may contribute to delayed improvement and increase the risk of death. The study hypothesizes that use of inhaled corticosteroids in addition to standard treatment in children hospitalized with ALRI will be associated with reduced morbidity and mortality and that the improvement will be more marked in children diagnosed with asthma posthoc. Outcomes: Reduction in case fatality, Time to normalization of respiratory rate, Time to normalization of oxygen saturation, Duration of hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 to 59 months with cough and or difficult breathing

Exclusion Criteria:

* Presence of a serious concurrent illness such as meningitis, Children with congenital or acquired heart disease Severe anaemia Measles pneumonia Foreign body inhalation A confirmed diagnosis of pulmonary tuberculosis

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1010 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
case fatality | In-hospital mortality
  Proportion of enrolled children who die of severe acute lower respiratory infection in the intervention compared to the placebo

SECONDARY OUTCOMES:
Hospital stay | From admission to discharge
  The average duration of hospitalisation in the intervention compared to the placebo group. The average duration of hospitalisation in the pneumonia compared to the children with asthma per treatment arm.

OTHER OUTCOMES:
Health workers' attitudes and perceptions towards use of inhaled corticosteroids, Mothers/ caretakers' level of satisfaction with the treatment | study period
  Proportion of health workers who know how to treat ALRI in children, attitudes and perceptions towards use of inhaled corticosteroids Mothers/ caretakers' level of satisfaction with the treatment given during hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Ndeezi, PhD, Principal Investigator — Makerere University; Marianne S Østergaard, PhD, Study Chair — University of Copenhagen; James K Tumwine, PhD, Study Director — Makerere University
Locations (1):
- Makerere University College of Health Sciences, Kampala, Uganda

REFERENCES:
- [Background] Ostergaard MS, Nantanda R, Tumwine JK, Aabenhus R. Childhood asthma in low income countries: an invisible killer? Prim Care Respir J. 2012 Jun;21(2):214-9. doi: 10.4104/pcrj.2012.00038. PMID 22623048
- [Background] Ostergaard MS, Prahl P. Diagnosis of preschool asthma: parents' comments and typical phrases may ease history-taking. Prim Care Respir J. 2007 Jun;16(3):194-5. doi: 10.3132/pcrj.2007.00035. No abstract available. PMID 17530145
- [Background] Sachdev HP, Mahajan SC, Garg A. Improving antibiotic and bronchodilator prescription in children presenting with difficult breathing: experience from an urban hospital in India. Indian Pediatr. 2001 Aug;38(8):827-38. PMID 11520993
- [Background] Okoromah CN, Oviawe O. Is childhood asthma underdiagnosed and undertreated? Niger Postgrad Med J. 2002 Dec;9(4):221-5. PMID 12690683
- [Background] Nantanda R, Hildenwall H, Peterson S, Kaddu-Mulindwa D, Kalyesubula I, Tumwine JK. Bacterial aetiology and outcome in children with severe pneumonia in Uganda. Ann Trop Paediatr. 2008 Dec;28(4):253-60. doi: 10.1179/146532808X375404. PMID 19021940
- See also: PUBMED — http://www.ncbi.nlm.nih.gov/pubmed/17710485